CLINICAL TRIAL: NCT01429610
Title: Phase 2 Study Evaluating the Efficacy of Rituximab Plus Modified VPDL for Newly Diagnosed CD20-Positive Adult Acute Lymphoblastic Leukemia
Brief Title: Rituximab+mVPDL for CD20(+) Adult Acute Lymphoblastic Leukemia
Acronym: RADICAL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Je-Hwan Lee, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KALLA0804
Record Dates: First submitted 2011-08-30; First posted 2011-09-07 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Precursor Cell Lymphoblastic Leukemia-Lymphoma
Keywords: acute lymphoblastic leukemia; rituximab; VPDL; CD20
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Rituximab; Asparaginase; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab+mVPDL (Experimental): Patients who were CD20(+), newly-diagnosed adult ALL and treated with rituximab + mVPDL treatment plan
  Interventions: Drug: Rituximab+mVPDL

INTERVENTIONS:
Drug: Rituximab+mVPDL — 1. Induction:
     * Dauno 90 mg/m2/d by civ (d1-3)
     * Vinc 2 mg iv (d1, 8)
     * Pred 60 mg/m2/d po (d1-14)
     * for Ph(-): L-asp 4,000 units/m2/day im/sc (d17-28) for Ph(+): Imatinib 600mg/d po qd (d8-continue till the end of maintenance or just before alloHCT)
     * Rituximab 375mg/m2/d (d8)
  2. Consolidation A (cycle1)
     * D 45 mg/m2/day by continuous iv (d1, 2)
     * V 2 mg iv (d1, 8)
     * P 60 mg/m2/day po (d1-14)
     * for Ph(-): L-asp (d1-14) for Ph(+): Imatinib
     * Rituximab 375mg/m2/d (d8)
  3. Consolidation B (cycles2&4)
     * Cyt 2,000 mg/m2/d iv over 2 hr (d1-4)
     * Eto 150 mg/m2/d iv over 3 hr (d1-4)
     * Rituximab 375mg/m2/d d8
  4. Consolidation C (cycles 3&5)
     * Methotrexate 220 mg/m2 iv bolus, then 60mg/m2/h for 36 hr (d1-2, 15-16)
     * Leucovorin 50 mg/m2 iv every 6hr for 3 doses,
     * Rituximab 375mg/m2/d (d8&22)
  5. Maintenance (for 2 years)
     - for Ph(-): 6- Mercaptopurine 60 mg/m2 po qd Methotrexate 20 mg/m2 po qw for Ph(+): imatinib 600mg/d po qd
  6. Consider alloHCT
  Other Names: Mabthera; VCS; Daunobrastina; Solondo; Leunase; Cytarabine; Efosin; DBLMethotrexate

SUMMARY:
The investigators would like to propose a phase-2 prospective multicenter trial evaluating the efficacy of rituximab combination with our current chemotherapy strategy for adult Acute Lymphoblastic Leukemia (ALL), in order to prove out whether the addition of rituximab during induction, consolidation, and post-alloHCT status can improve the outcome in terms of relapse-free survival (RFS) when compared with our prior data as a historical control.

DETAILED DESCRIPTION:
According to the recent results on the outcome of escalated daunorubicin-based protocol for adult ALL which has been performed by 'Adult ALL Working Party of the Korean Society of Hematology' (data were announced at 2010 Annual Meeting of ASCO, Chicago, IL), CR rate of 90.6% was satisfactory, but the 2-year / 3-year disease-free survival (DFS) were disappointing (43.6% and 39.9%, respectively), which means that the adequate post-remission therapy to control minimal residual disease after the achievement of CR is very important to improve the outcome of adult ALL.

Allogeneic hematopoietic cell transplantation (AlloHCT) is recommended as a post-remission therapy for patients with adult ALL, and reduced intensity conditioning has been tried to decrease TRM rate. However, many patients received consolidation chemotherapy rather than alloHCT owing to the absence of HLA-matched donor, limitation of age, and combined comorbidities (among 190 patients who have been included in our previously-mentioned study, only 52.3% received alloHCT).

Recently, stagnation in the treatment of adult ALL appears to be reached, maybe due to a borderline for further intensification of chemotherapeutic dose. Dose-escalation strategy has many difficulties in adoption for the treatment of adult ALL in terms of increased morbidity and mortality, not to mention the efficacy of such strategies. New, preferably non-chemotherapy approaches (maybe targeted therapy) are therefore urgently required.

For Ph(+) ALL, the introduction of BCR/ABL tyrosine kinase inhibitor has improved the treatment outcome with tolerable toxicities. Applying a similar strategy to Ph(-) ALL, targeting leukemia surface antigens with monoclonal antibodies is another promising strategy.

CD 20 expression of at least 20% has been known to be found in 22-48% of pre-B ALL, and appears to be associated with a poor prognosis, although there are controversies in pediatric patients. Based on the significant improvement of the outcome in B-cell NHL, preliminary data regarding the use of rituximab in frontline therapy for CD20-positive precursor B-cell ALL suggest its use may be beneficial. Especially, monoclonal antibodies are thought to be more effective when combined with chemotherapy and treated in the state of minimal residual disease, which suggests the interest of evaluating rituximab combined to current chemotherapy of adult ALL. Recent data on the efficacy of rituximab-combined chemotherapy showed that rates of CR and OS were superior with the modified hyperCVAD and rituximab regimens compared with standard hyper-CVAD (70% versus 38%, p<0.001) in younger (age < 60 years) CD20-positive subset, although it was an analysis of different patient groups who were treated with various regimen5.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were previously untreated and had either ALL or high-risk lymphoblastic lymphoma.
* Patients whose leukemic blast cells express ≥20% of CD20 antigens at time of diagnosis
* No prior chemotherapy for leukemia (use of hydroxyurea or leukapheresis are permitted.)
* Estimated life expectancy of more than 3 months
* ECOG performance status of 2 or lower, Karnofsky scale > 60
* Adequate cardiac function (EF>45%) on echocardiogram or Heart scan (MUGA scan)
* 15 years of age and over.
* Adequate renal function (creatinine<1.5 mg/dL)
* Adequate hepatic function. (Bilirubin<1.5 mg/dL, transaminases levels<3 times the upper normal limit [5 times for patients with liver metastasis or hepatomegaly]). Even the initial level exceed the upper limits, patient will be acceptable when the levels on day 8 satisfies the inclusion criteria.
* All patients gave written informed consent according to guidelines at each institution's committee on human research.

Exclusion Criteria:

* Acute biphenotypic leukemia, acute biclonal leukemia, or acute mixed leukemia
* Presence of significant uncontrolled active infection
* Presence of uncontrolled bleeding
* Any coexisting major illness or organ failure
* Patients with psychiatric disorder or mental deficiency severe as to make compliance with the treatment unlike, and making informed consent impossible
* Nursing women, pregnant women, women of childbearing potential who do not want adequate contraception
* Patients with a diagnosis of prior malignancy unless disease-free for at least 5 years following therapy with curative intent (except curatively treated nonmelanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-11; Primary Completion 2018-01-01 (Actual); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
relapse-free survival (RFS) rate | 2 years

SECONDARY OUTCOMES:
complete remission (CR) rates | 4 weeks (from the initiation of induction treatment)
  among total patients / each subset of subsets A.
  [Subset A]
  1. Precursor B-cell vs. T-cell
  2. Younger (age<60 years) vs. older (age≥60 years)
  3. Risk group: standard vs. high
relapse-free survival rates | 2 years
  among patients in each subset of A & B.
  [Subset A]
  1. Precursor B-cell vs. T-cell
  2. Younger (age<60 years) vs. older (age≥60 years)
  3. Risk group: standard vs. high.
     [Subset B]
  4. AlloHCT recipients vs. non-recipients.
overall survival rates | 2 years
  among total patients / each subset of A & B
  [Subset A]
  1. Precursor B-cell vs. T-cell
  2. Younger (age<60 years) vs. older (age≥60 years)
  3. Risk group: standard vs. high [Subset B]
  4. AlloHCT recipients vs. non-recipients.
Cumulative incidence and maximal severity of acute / chronic graft-versus-host disease | 2 years
  among alloHCT recipients

CONTACTS AND LOCATIONS:
Overall Officials: Young Don Joo, MD, PhD, Principal Investigator — Inje University Haeundae Paik Hospital
Locations (19):
- South Korea (19):
  - Chonnam National University Hwasun Hospital, Hwasun, Chollanamdo
  - Hematologic Oncology Clinic, National Cancer Center, Ilsan, Kongki
  - Division of Hematology-Oncology, Dong-A University College of Medicine, Busan
  - Dong-A University College of Medicine, Busan
  - Inje University Busan Paik Hospital, Busan
  - Inje University Haeundae-Paik Hospital, Busan
  - Kosin University College of Medicine, Kosin University Gospel Hospital, Busan
  - Catholic University of Daegu School of Medicine, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National Unviersity Hospital, Daegu
  - Yeungnam University College of Medicine, Daegu
  - Chungnam National University Hospital, Daejeon
  - Asan Medical Center, University of Ulsan College of Medicine, Seoul
  - Chung-Ang University Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Soonchunhyang University Hospital, Seoul
  - Ulsan University Hospital, University of Ulsan College of Medicine, Ulsan

REFERENCES:
- [Background] Boissel N, Auclerc MF, Lheritier V, Perel Y, Thomas X, Leblanc T, Rousselot P, Cayuela JM, Gabert J, Fegueux N, Piguet C, Huguet-Rigal F, Berthou C, Boiron JM, Pautas C, Michel G, Fiere D, Leverger G, Dombret H, Baruchel A. Should adolescents with acute lymphoblastic leukemia be treated as old children or young adults? Comparison of the French FRALLE-93 and LALA-94 trials. J Clin Oncol. 2003 Mar 1;21(5):774-80. doi: 10.1200/JCO.2003.02.053. Epub 2003 Mar 1. PMID 12610173
- [Background] Hallbook H, Gustafsson G, Smedmyr B, Soderhall S, Heyman M; Swedish Adult Acute Lymphocytic Leukemia Group; Swedish Childhood Leukemia Group. Treatment outcome in young adults and children >10 years of age with acute lymphoblastic leukemia in Sweden: a comparison between a pediatric protocol and an adult protocol. Cancer. 2006 Oct 1;107(7):1551-61. doi: 10.1002/cncr.22189. PMID 16955505
- [Background] Todeschini G, Tecchio C, Meneghini V, Pizzolo G, Veneri D, Zanotti R, Ricetti MM, Solero P, April F, Perona G. Estimated 6-year event-free survival of 55% in 60 consecutive adult acute lymphoblastic leukemia patients treated with an intensive phase II protocol based on high induction dose of daunorubicin. Leukemia. 1998 Feb;12(2):144-9. doi: 10.1038/sj.leu.2400912. PMID 9519775
- [Background] Thomas D, O'Brien S, Faderl S, Ravandi F, Jabbour E, Pierce S, Cortes J, Kantarjian H. Anthracycline dose intensification in adult acute lymphoblastic leukemia: lack of benefit in the context of the fractionated cyclophosphamide, vincristine, doxorubicin, and dexamethasone regimen. Cancer. 2010 Oct 1;116(19):4580-9. doi: 10.1002/cncr.25319. PMID 20572037
- [Background] Tomblyn MB, Arora M, Baker KS, Blazar BR, Brunstein CG, Burns LJ, DeFor TE, Dusenbery KE, Kaufman DS, Kersey JH, MacMillan ML, McGlave PB, Miller JS, Orchard PJ, Slungaard A, Tomblyn MR, Vercellotti GM, Verneris MR, Wagner JE, Weisdorf DJ. Myeloablative hematopoietic cell transplantation for acute lymphoblastic leukemia: analysis of graft sources and long-term outcome. J Clin Oncol. 2009 Aug 1;27(22):3634-41. doi: 10.1200/JCO.2008.20.2960. Epub 2009 Jul 6. PMID 19581540
- [Background] Bachanova V, Verneris MR, DeFor T, Brunstein CG, Weisdorf DJ. Prolonged survival in adults with acute lymphoblastic leukemia after reduced-intensity conditioning with cord blood or sibling donor transplantation. Blood. 2009 Mar 26;113(13):2902-5. doi: 10.1182/blood-2008-10-184093. Epub 2009 Jan 28. PMID 19179301
- [Background] Goldstone AH, Richards SM, Lazarus HM, Tallman MS, Buck G, Fielding AK, Burnett AK, Chopra R, Wiernik PH, Foroni L, Paietta E, Litzow MR, Marks DI, Durrant J, McMillan A, Franklin IM, Luger S, Ciobanu N, Rowe JM. In adults with standard-risk acute lymphoblastic leukemia, the greatest benefit is achieved from a matched sibling allogeneic transplantation in first complete remission, and an autologous transplantation is less effective than conventional consolidation/maintenance chemotherapy in all patients: final results of the International ALL Trial (MRC UKALL XII/ECOG E2993). Blood. 2008 Feb 15;111(4):1827-33. doi: 10.1182/blood-2007-10-116582. Epub 2007 Nov 29. PMID 18048644
- [Background] Pituch-Noworolska A, Hajto B, Mazur B, Sonta-Jakimczyk D, Balwierz W, Janota-Krawczyk E, Kowalska H, Malinowska I, Modzelewska M, Wasik M. Expression of CD20 on acute lymphoblastic leukemia cells in children. Neoplasma. 2001;48(3):182-7. PMID 11583286
- [Background] Maury S, Huguet F, Leguay T, Lacombe F, Maynadie M, Girard S, de Labarthe A, Kuhlein E, Raffoux E, Thomas X, Chevallier P, Buzyn A, Delannoy A, Chalandon Y, Vernant JP, Rousselot P, Macintyre E, Ifrah N, Dombret H, Bene MC; Group for Research on Adult Acute Lymphoblastic Leukemia. Adverse prognostic significance of CD20 expression in adults with Philadelphia chromosome-negative B-cell precursor acute lymphoblastic leukemia. Haematologica. 2010 Feb;95(2):324-8. doi: 10.3324/haematol.2009.010306. Epub 2009 Sep 22. PMID 19773266
- [Background] Borowitz MJ, Shuster J, Carroll AJ, Nash M, Look AT, Camitta B, Mahoney D, Lauer SJ, Pullen DJ. Prognostic significance of fluorescence intensity of surface marker expression in childhood B-precursor acute lymphoblastic leukemia. A Pediatric Oncology Group Study. Blood. 1997 Jun 1;89(11):3960-6. PMID 9166833
- [Background] Jeha S, Behm F, Pei D, Sandlund JT, Ribeiro RC, Razzouk BI, Rubnitz JE, Hijiya N, Howard SC, Cheng C, Pui CH. Prognostic significance of CD20 expression in childhood B-cell precursor acute lymphoblastic leukemia. Blood. 2006 Nov 15;108(10):3302-4. doi: 10.1182/blood-2006-04-016709. Epub 2006 Aug 8. PMID 16896151
- [Background] Thomas DA, O'Brien S, Jorgensen JL, Cortes J, Faderl S, Garcia-Manero G, Verstovsek S, Koller C, Pierce S, Huh Y, Wierda W, Keating MJ, Kantarjian HM. Prognostic significance of CD20 expression in adults with de novo precursor B-lineage acute lymphoblastic leukemia. Blood. 2009 Jun 18;113(25):6330-7. doi: 10.1182/blood-2008-04-151860. Epub 2008 Aug 14. PMID 18703706
- [Background] Al Gwaiz LA, Bassioni W. Immunophenotyping of acute lymphoblastic leukemia using immunohistochemistry in bone marrow biopsy specimens. Histol Histopathol. 2008 Oct;23(10):1223-8. doi: 10.14670/HH-23.1223. PMID 18712674
- [Background] Claviez A, Eckert C, Seeger K, Schrauder A, Schrappe M, Henze G, von Stackelberg A. Rituximab plus chemotherapy in children with relapsed or refractory CD20-positive B-cell precursor acute lymphoblastic leukemia. Haematologica. 2006 Feb;91(2):272-3. PMID 16461321
- [Background] Thomas DA, Faderl S, O'Brien S, Bueso-Ramos C, Cortes J, Garcia-Manero G, Giles FJ, Verstovsek S, Wierda WG, Pierce SA, Shan J, Brandt M, Hagemeister FB, Keating MJ, Cabanillas F, Kantarjian H. Chemoimmunotherapy with hyper-CVAD plus rituximab for the treatment of adult Burkitt and Burkitt-type lymphoma or acute lymphoblastic leukemia. Cancer. 2006 Apr 1;106(7):1569-80. doi: 10.1002/cncr.21776. PMID 16502413
- [Background] Thomas DA, O'Brien S, Faderl S, Garcia-Manero G, Ferrajoli A, Wierda W, Ravandi F, Verstovsek S, Jorgensen JL, Bueso-Ramos C, Andreeff M, Pierce S, Garris R, Keating MJ, Cortes J, Kantarjian HM. Chemoimmunotherapy with a modified hyper-CVAD and rituximab regimen improves outcome in de novo Philadelphia chromosome-negative precursor B-lineage acute lymphoblastic leukemia. J Clin Oncol. 2010 Aug 20;28(24):3880-9. doi: 10.1200/JCO.2009.26.9456. Epub 2010 Jul 26. PMID 20660823
- [Background] Coiffier B, Lepage E, Briere J, Herbrecht R, Tilly H, Bouabdallah R, Morel P, Van Den Neste E, Salles G, Gaulard P, Reyes F, Lederlin P, Gisselbrecht C. CHOP chemotherapy plus rituximab compared with CHOP alone in elderly patients with diffuse large-B-cell lymphoma. N Engl J Med. 2002 Jan 24;346(4):235-42. doi: 10.1056/NEJMoa011795. PMID 11807147
- [Background] Feugier P, Van Hoof A, Sebban C, Solal-Celigny P, Bouabdallah R, Ferme C, Christian B, Lepage E, Tilly H, Morschhauser F, Gaulard P, Salles G, Bosly A, Gisselbrecht C, Reyes F, Coiffier B. Long-term results of the R-CHOP study in the treatment of elderly patients with diffuse large B-cell lymphoma: a study by the Groupe d'Etude des Lymphomes de l'Adulte. J Clin Oncol. 2005 Jun 20;23(18):4117-26. doi: 10.1200/JCO.2005.09.131. Epub 2005 May 2. PMID 15867204
- [Background] Hiddemann W, Kneba M, Dreyling M, Schmitz N, Lengfelder E, Schmits R, Reiser M, Metzner B, Harder H, Hegewisch-Becker S, Fischer T, Kropff M, Reis HE, Freund M, Wormann B, Fuchs R, Planker M, Schimke J, Eimermacher H, Trumper L, Aldaoud A, Parwaresch R, Unterhalt M. Frontline therapy with rituximab added to the combination of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) significantly improves the outcome for patients with advanced-stage follicular lymphoma compared with therapy with CHOP alone: results of a prospective randomized study of the German Low-Grade Lymphoma Study Group. Blood. 2005 Dec 1;106(12):3725-32. doi: 10.1182/blood-2005-01-0016. Epub 2005 Aug 25. PMID 16123223
- [Background] Griffin TC, Weitzman S, Weinstein H, Chang M, Cairo M, Hutchison R, Shiramizu B, Wiley J, Woods D, Barnich M, Gross TG; Children's Oncology Group. A study of rituximab and ifosfamide, carboplatin, and etoposide chemotherapy in children with recurrent/refractory B-cell (CD20+) non-Hodgkin lymphoma and mature B-cell acute lymphoblastic leukemia: a report from the Children's Oncology Group. Pediatr Blood Cancer. 2009 Feb;52(2):177-81. doi: 10.1002/pbc.21753. PMID 18816698
- [Background] Hallek M, Fischer K, Fingerle-Rowson G, Fink AM, Busch R, Mayer J, Hensel M, Hopfinger G, Hess G, von Grunhagen U, Bergmann M, Catalano J, Zinzani PL, Caligaris-Cappio F, Seymour JF, Berrebi A, Jager U, Cazin B, Trneny M, Westermann A, Wendtner CM, Eichhorst BF, Staib P, Buhler A, Winkler D, Zenz T, Bottcher S, Ritgen M, Mendila M, Kneba M, Dohner H, Stilgenbauer S; International Group of Investigators; German Chronic Lymphocytic Leukaemia Study Group. Addition of rituximab to fludarabine and cyclophosphamide in patients with chronic lymphocytic leukaemia: a randomised, open-label, phase 3 trial. Lancet. 2010 Oct 2;376(9747):1164-74. doi: 10.1016/S0140-6736(10)61381-5. PMID 20888994
- [Background] Ratanatharathorn V, Pavletic S, Uberti JP. Clinical applications of rituximab in allogeneic stem cell transplantation: anti-tumor and immunomodulatory effects. Cancer Treat Rev. 2009 Dec;35(8):653-61. doi: 10.1016/j.ctrv.2009.07.004. Epub 2009 Aug 13. PMID 19682801
- [Background] Dworzak MN, Schumich A, Printz D, Potschger U, Husak Z, Attarbaschi A, Basso G, Gaipa G, Ratei R, Mann G, Gadner H. CD20 up-regulation in pediatric B-cell precursor acute lymphoblastic leukemia during induction treatment: setting the stage for anti-CD20 directed immunotherapy. Blood. 2008 Nov 15;112(10):3982-8. doi: 10.1182/blood-2008-06-164129. Epub 2008 Sep 9. PMID 18780832
- [Background] Stanciu-Herrera C, Morgan C, Herrera L. Anti-CD19 and anti-CD22 monoclonal antibodies increase the effectiveness of chemotherapy in Pre-B acute lymphoblastic leukemia cell lines. Leuk Res. 2008 Apr;32(4):625-32. doi: 10.1016/j.leukres.2007.07.002. Epub 2007 Aug 15. PMID 17706771
- [Background] Gaipa G, Basso G, Maglia O, Leoni V, Faini A, Cazzaniga G, Bugarin C, Veltroni M, Michelotto B, Ratei R, Coliva T, Valsecchi MG, Biondi A, Dworzak MN; I-BFM-ALL-FCM-MRD Study Group. Drug-induced immunophenotypic modulation in childhood ALL: implications for minimal residual disease detection. Leukemia. 2005 Jan;19(1):49-56. doi: 10.1038/sj.leu.2403559. PMID 15538405
- [Background] Gokbuget N, Hoelzer D. Treatment with monoclonal antibodies in acute lymphoblastic leukemia: current knowledge and future prospects. Ann Hematol. 2004 Apr;83(4):201-5. doi: 10.1007/s00277-003-0752-8. Epub 2003 Nov 26. PMID 14648023
- [Background] Bachanova V, Sandhu K, Yohe S, Cao Q, Burke MJ, Verneris MR, Weisdorf D. Allogeneic hematopoietic stem cell transplantation overcomes the adverse prognostic impact of CD20 expression in acute lymphoblastic leukemia. Blood. 2011 May 12;117(19):5261-3. doi: 10.1182/blood-2011-01-329573. Epub 2011 Mar 14. PMID 21403127
- [Background] Cutler C, Miklos D, Kim HT, Treister N, Woo SB, Bienfang D, Klickstein LB, Levin J, Miller K, Reynolds C, Macdonell R, Pasek M, Lee SJ, Ho V, Soiffer R, Antin JH, Ritz J, Alyea E. Rituximab for steroid-refractory chronic graft-versus-host disease. Blood. 2006 Jul 15;108(2):756-62. doi: 10.1182/blood-2006-01-0233. Epub 2006 Mar 21. PMID 16551963
- [Background] Mohty M, Marchetti N, El-Cheikh J, Faucher C, Furst S, Blaise D. Rituximab as salvage therapy for refractory chronic GVHD. Bone Marrow Transplant. 2008 May;41(10):909-11. doi: 10.1038/bmt.2008.12. Epub 2008 Feb 18. No abstract available. PMID 18278073
- [Background] Okamoto M, Okano A, Akamatsu S, Ashihara E, Inaba T, Takenaka H, Katoh N, Kishimoto S, Shimazaki C. Rituximab is effective for steroid-refractory sclerodermatous chronic graft-versus-host disease. Leukemia. 2006 Jan;20(1):172-3. doi: 10.1038/sj.leu.2403996. No abstract available. PMID 16239908
- [Background] Zaja F, Bacigalupo A, Patriarca F, Stanzani M, Van Lint MT, Fili C, Scime R, Milone G, Falda M, Vener C, Laszlo D, Alessandrino PE, Narni F, Sica S, Olivieri A, Sperotto A, Bosi A, Bonifazi F, Fanin R; GITMO (Gruppo Italiano Trapianto Midollo Osseo). Treatment of refractory chronic GVHD with rituximab: a GITMO study. Bone Marrow Transplant. 2007 Aug;40(3):273-7. doi: 10.1038/sj.bmt.1705725. Epub 2007 Jun 4. PMID 17549053
- [Background] Kebriaei P, Saliba RM, Ma C, Ippoliti C, Couriel DR, de Lima M, Giralt S, Qazilbash MH, Gajewski JL, Ha CS, Champlin RE, Khouri IF. Allogeneic hematopoietic stem cell transplantation after rituximab-containing myeloablative preparative regimen for acute lymphoblastic leukemia. Bone Marrow Transplant. 2006 Aug;38(3):203-9. doi: 10.1038/sj.bmt.1705425. Epub 2006 Jun 26. PMID 16799614
- [Derived] Baek DW, Park HS, Sohn SK, Kim DY, Kim I, Ahn JS, Do YR, Lee SR, Eom HS, Lee WS, Kim SH, Lee HS, Lee YJ, Moon JH, Lee JH; Adult Acute Lymphoblastic Leukemia Working Party, the Korean Society of Hematology. Rituximab plus multiagent chemotherapy for newly diagnosed CD20-positive acute lymphoblastic leukemia: a prospective phase II study. Korean J Intern Med. 2023 Sep;38(5):734-746. doi: 10.3904/kjim.2022.401. Epub 2023 Jun 20. PMID 37334511